CLINICAL TRIAL: NCT05402787
Title: The Effect of Virtual Visit to Mothers With Infants in the Neonatal Intensive Care Unit on Mothers' Attachment and Satisfaction
Brief Title: Impact of Virtual Visit on Mothers' Attachment and Satisfaction
Acronym: Virtualvisit
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sakarya University (Other)
Responsible Party: Principal Investigator, dilek menekşe, Assistant professor, Sakarya University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: E-16214662-050.01.04-6777-02
Record Dates: First submitted 2022-04-08; First posted 2022-06-02 (Actual); Last update posted 2022-06-02 (Actual); Status verified 2022-05

CONDITIONS: Virtual; Attachment; Satisfaction
Keywords: Virtual visit; Attachment; Satisfaction; Newborn
MeSH Terms: conditions — Personal Satisfaction

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Trial
Who Masked: Outcomes Assessor
Masking Description: Single-blind (researchers are not blinded) randomization will be provided as the virtual visitation to mothers will be implemented by researchers. The statistician was also blinded for the data analysis purpose
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): The virtual visit will be started within the first 24 hours after birth. Mothers in this group will be informed about how the virtual visit will be. The virtual visit will be made online through the Whatshup video call program. The virtual visit will be twice a day, starting 24 hours after birth until the baby's first meeting with the mother. The first virtual visit to be made during the day will be aimed at understanding the mother's feelings, increasing her motivation and informing about the clinical condition of the baby. In the second interview, it will be supported to provide approximately 10 minutes of visual and audio communication that will help the mother to establish a connection with her baby. During the virtual visiting hour, the videos of the baby will be sent to the mother so that the mother can watch it. In each visit, it will be ensured that the mother sees her baby in every situation by paying attention to the fact that the baby is in a different situation.
  Interventions: Other: Virtual visit
- Control Groups (No Intervention): The mothers in the control group will be followed in line with the hospital's routine health monitoring and information.

INTERVENTIONS:
Other: Virtual visit — A virtual visit will be made to mothers whose babies are hospitalized in the neonatal intensive care unit
  Arms: Experimental

SUMMARY:
Virtual visit, which is frequently used in the field of health in line with the latest technological developments, is accepted as a unique opportunity that allows babies and their families to connect in real time. Studies have reported that virtual visits increase mothers' sense of closeness to their babies and have positive effects on the attachment process (Dunham and Marin 2020; Flacking et al. 2014; Joshi et al. 2016). It is clearly emphasized that healthy and securely attached babies have positive effects on health. This study was designed as a randomized controlled experimental study in order to determine the effect of virtual visit applied to mothers whose babies are in the neonatal intensive care unit on their attachment and satisfaction.

Research Hypotheses:

H0: There is no difference between the attachment and satisfaction of mothers whose babies were hospitalized in the neonatal intensive care unit, and those who did not receive virtual visits.

H1: Attachment and satisfaction of mothers whose babies are hospitalized in the neonatal intensive care unit with virtual visits are higher than mothers who do not receive virtual visits.

DETAILED DESCRIPTION:
In recent years, studies on parent-infant bonding, which have an impact on child health and affect the entire life of the child, have been continuing increasingly. Attachment refers to a mutual, warm, loving and secure attachment relationship. Attachment, which is an important concept in the development process of human beings (Güleç and Kavak 2013; Çınar and Köse 2015). It is a simultaneous and continuous process that starts in the prenatal period and develops gradually in the birth and postnatal period (Köse et al. 2013). In the postpartum period, the rapid and safe interaction between the mother and the baby and meeting the needs of the baby make attachment stronger. People who have developed a sense of trust and experienced a secure relationship and attachment process, especially during infancy, can be in a more advantageous position in terms of healthy growth, character development and mental health (Menekşe and Çınar 2020). In addition, the attachment of the mother to her baby with love is important in the development of parental identity and adaptation to the role of the mother. While providing the care of the baby by the mother gives happiness and pleasure to the mother along with the sense of competence, the baby encodes some mental and motivational representations towards the caregiver (Mercer 2004; Nacar and Gökkaya 2019). In some cases, this process may be adversely affected in the postpartum period. One of the factors that negatively affect the mother-infant interaction process is prematurity and hospitalization of the baby in the neonatal intensive care unit. (Jobs 2007).

According to the results of the Turkey Demographic and Health Survey (2018), the rate of low birth weight babies in Turkey is 12%. Babies born prematurely or hospitalized in the neonatal intensive care unit due to a disease spend the first days and even the first months of their lives receiving intensive medical treatment and care . Premature babies in pediatrics are included in the patient group with the longest hospital stay. In this case, parents may experience complex emotions such as shock, anxiety, grief, denial, hopelessness, anger, inadequacy and self-confidence (Pisoni et al. 2014b; İşler 2007; Öztürk and Saruhan 2013; Flacking et al. 2014). Premature births, which are a stressful experience with long-term effects for families, affect maternal attachment characteristics and process (Guex et al. 2011). Reasons such as the birth being before the expected date, the transfer of the baby to the neonatal intensive care unit due to different than imagined or health problems, the fear of losing the baby, the inability to interact with the baby or not being able to see at all, insufficient information about the baby's problems, the mother's discharge by leaving the baby in the hospital. affects the relationship negatively (İşler 2007; Scatliffe et l. 2019). Therefore, alongside the best possible medical treatment for the newborn, family-centered care plays a vital role in supporting parents and strengthening the parent-infant bond in these exceptional situations. Health professionals should contribute to parent-infant bonding by creating an opportunity to be with their children by encouraging parents to observe, talk, touch, provide skin-to-skin contact and participate in care in the neonatal intensive care unit.

Virtual visit, which is frequently used in the field of health in line with the latest technological developments, is accepted as a unique opportunity that allows babies and their families to connect in real time. Studies have reported that virtual visitation has increased mothers' sense of closeness to their babies and has positive effects on the attachment process (Dunham and Marin 2020; Flacking et al. 2014; Joshi et al. 2016). In addition, virtual visits are used to keep both healthcare staff and families safe during the coronavirus outbreak. The implementation of visits is also advantageous in terms of being simple and cost-effective.In this extraordinary period, which we have been experiencing with the COVID-19 pandemic, which has deeply affected the world, some decisions are taken on the basis of country and institution-based visits, in order to protect the vulnerable group of premature babies from this infection. Although these decisions create physical barriers to attachment, such as the family's inability to see and interact with their baby, this situation can be difficult, frightening and sometimes traumatic for the family who is emotionally distant from their baby. Expressing the feelings of families with babies in intensive care, maintaining their interaction with their baby, and ensuring the continuity of breastfeeding and care trainings in line with the needs of the family through virtual visits has once again revealed the necessity.

In the light of this information; The aim of this study was to determine the effect of the virtual visit applied to the mothers whose babies are in the neonatal intensive care unit on their attachment and satisfaction.

Method: This research is a randomized controlled experimental study. The sample of the research was collected between May 2022 and May 2023 in T.C. Ministry of Health Sakarya Provincial Health Directorate Sakarya Training and Research Hospital Gynecology and Pediatrics Service Building in the neonatal intensive care unit, 32-34. Mothers of premature babies born primiparly in the week of gestation will form. Power analysis was performed using the G*Power (v3.1.7) program to determine the number of samples (Faul, Erdfelder, Buchner and Lang 2013). The effect width value was taken as 0.70 as the method used in cases where it is not known how many units the difference is important between the groups. The effect width value of 0.20 is very high, 0.50 is medium, and 0.80 is below the maximum acceptance constraint. The higher the power of the study, the more precise the measurement is in finding the difference. The power is expected to be 0.80 and above. However, some experts emphasize that this limit is between 0.70 and 0.90. In case the probability of type 1 error (α) was 0.05 (95% confidence level), 80% power level, and the effect width value was 0.70, the study was planned with the mothers of a total of 68 premature babies, 34 babies for each group. In the study, a total of 68 mothers forming the sample will be divided into two groups as randomized controlled. The mothers to be assigned to the groups will be assigned through a computer-based random number generator program. The sample of the study will randomly allocated into two groups: a virtual visit to the intervention group, and the other group, which was the control group, will be followed by a routine visit of the service. Single-blind (researchers are not blinded) randomization will be provided since the virtual visit to mothers will be implemented by the researchers. The statistician was also blinded for the data analysis purpose. In the study, the data were collected from the "Mother Descriptive Information Form", "Preterm Descriptive Information Form", "Virtual Visit Follow-up Form" prepared by the researchers, "Maternal Attachment Scale" developed by Muller (1994) and validated by Kavlak Latour et al.( 2011) was developed by Latour et al. (2013), the short form of the scale was created by using the Empathic -30 questionnaire, which was validated by Tiryaki et al. (2020).

"Mother and Preterm Descriptive Information Form", "Maternal Attachment Scale" and "Empathic -30" scale will be filled in for mothers who agree to participate in the study before the first virtual visit 24 hours after birth. The virtual visit to the mothers in the experimental group will be applied twice a day, starting 24 hours after birth and until the baby's first meeting with the mother. The virtual visit will be made online through the Whatshup video call program. In addition to the routine visit of the clinic, the virtual visit will ensure the continuity of the mother's communication with her baby. The data will be recorded in the Virtual Visit Tracking Form. The mothers in the control group will be followed in line with the hospital's routine health monitoring and information.

At the baby's discharge, they will be asked to fill in the Maternal Attachment Scale and Empathic -30 scale, and one month after the discharge, the Maternal Attachment Scale will be filled with the online questionnaire method by sending a URL address link to their e-mail/ WhatsApp. In the evaluation of data, statistical analyzes will be performed using the SPSS package program. The Kolmogorov-Smirnov (K-S) test will be used for normality. In order to determine whether there is a difference in the dependent variables compared to independent variables, the independent group t-test will be used if the distribution is normal in independent variables with two options, and Mann Whitney-U test will be used if distribution is not normal. The results will be evaluated at a confidence level of 95% and at a level of significance of p<0.05.

ELIGIBILITY:
Inclusion Criteria:

* • Premature (>32 and and <35 GW) of the newborn

  * To be admitted to the neonatal intensive care unit within the first 24 hours after birth
  * Absence of visible congenital anomaly (Cleft palate, cleft lip, craniofacial anomaly such as facial muscle paralysis etc.)
  * Hospitalization of the newborn in the neonatal intensive care unit for at least 1 week and the continuation of the virtual visit
  * Absence of a diagnosed psychiatric history of the mother
  * Mother's willingness to participate in the study
  * The mother has a primiparous and singleton baby
  * Mother is over 18 years old
  * The mother can speak and understand Turkish well and be literate
  * Pregnancy not realized by assisted reproductive technique
  * The mother who has a smart phone, computer, tablet and wireless internet will be included in the study.

Exclusion Criteria:

* • Premature (<32 and >35 GW) of the newborn

  * Not being admitted to the neonatal intensive care unit within the first 24 hours after birth
  * Congenital anomaly in the newborn (Craniofacial anomaly such as cleft palate, cleft lip, paralysis of facial muscles)
  * Discharge of the newborn before 1 week
  * Mother's unwillingness to participate in the study
  * Mother's illiteracy
  * The mother has a multiparous or multiple baby
  * The mother has a diagnosed psychiatric history
  * Mother is 18 years or younger
  * The mother did not have a smart phone, computer, tablet or wireless internet at the time of the study
  * Pregnancy with assisted reproductive technique
  * The mother's incomplete filling of the questionnaires

Ages: 19 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Mothers of infants hospitalized in the neonatal intensive care unit
Enrollment: 62 (Estimated)
Dates: Start 2022-06-20 (Estimated); Primary Completion 2022-06-20 (Estimated); Study Completion 2023-05-01 (Estimated)

PRIMARY OUTCOMES:
Evaluation of attachment in study and control groups | Change between attachment status before the first virtual visit (24 hours after birth), at least one week after admission to one month)., and one month after discharge.
  The Maternal Attachment Scale is a four-dimensional, one-dimensional, 26-item scale with each item ranging from 'always' to 'never'. Each item includes direct statements and always=4 points, often=3 points, sometimes=2 points. , is calculated as never = 1 point. The lowest score to be obtained from the scale is 26, and the highest score is 104. A high score indicates high maternal attachment.
Evaluation of family satisfaction in neonatal intensive care in study and control groups | Change between satisfaction before the first virtual visit (24 hours after birth) and at least one week after admission to one month
  The EMPATHIC-30 ((EMpowerment of Parents in THe Intensive Care ) scale is 6-point Likert-type (1= strongly disagree; 6 = strongly agree) and consists of five domains: knowledge (5 items), care and treatment (8 items) , organization (5 items), parent involvement (6 items) and professional attitude of staff (6 items) Scores ≤3 in each item are considered "Negative" while ≥4 points are considered "Positive" Average scores for each area ; (total score / total number of items in each field) formula

CONTACTS AND LOCATIONS:
Overall Officials: Dilek Menekşe, Asist. prof., Study Director — Sakarya University; Öznur Tiryaki, Asist. prof., Principal Investigator — Sakarya University; Nursan Çınar, Prof.Dr., Principal Investigator — Sakarya University; Seda Tecik, Res.Asist., Principal Investigator — Sakarya University; Hatice Solak, Nurse, Principal Investigator — Sakarya Training and Research Hospital; Meltem Karabay, Asist.Prof, Principal Investigator — Sakarya University; İbrahim Caner, Prof.Dr., Principal Investigator — Sakarya University

REFERENCES:
- [Background] Çınar N, Köse D. Aile -Bebek Bağlanma Süreci, Aile Temelli Sağlık Yaklaşımı, Ed: S.Kuğuoğlu, B.C. Demirbağ, 2015.
- [Background] Cinar N, Kose D, Altinkaynak S. The relationship between maternal attachment, perceived social support and breast-feeding sufficiency. J Coll Physicians Surg Pak. 2015 Apr;25(4):271-5. PMID 25899193
- [Background] Dunham MM, Marin T. NICU Maternal-Infant Bonding: Virtual Visitation as a Bonding Enhancement Tool. J Perinat Neonatal Nurs. 2020 Apr/Jun;34(2):171-177. doi: 10.1097/JPN.0000000000000484. PMID 32332447
- [Background] Flacking R, Lehtonen L, Thomson G, Axelin A, Ahlqvist S, Moran VH, Ewald U, Dykes F; Separation and Closeness Experiences in the Neonatal Environment (SCENE) group. Closeness and separation in neonatal intensive care. Acta Paediatr. 2012 Oct;101(10):1032-7. doi: 10.1111/j.1651-2227.2012.02787.x. Epub 2012 Aug 2. PMID 22812674
- [Background] Forcada-Guex M, Borghini A, Pierrehumbert B, Ansermet F, Muller-Nix C. Prematurity, maternal posttraumatic stress and consequences on the mother-infant relationship. Early Hum Dev. 2011 Jan;87(1):21-6. doi: 10.1016/j.earlhumdev.2010.09.006. Epub 2010 Oct 15. PMID 20951514
- [Background] İşler A. Prematüre bebeklerde anne-bebek ilişkisinin başlatılmasında yenidoğan hemşirelerinin rolü. Perinatoloji Dergisi 2007;15 (1): 1-6.
- [Background] Joshi A, Chyou PH, Tirmizi Z, Gross J. Web Camera Use in the Neonatal Intensive Care Unit: Impact on Nursing Workflow. Clin Med Res. 2016 Mar;14(1):1-6. doi: 10.3121/cmr.2015.1286. Epub 2016 Feb 10. PMID 26864509
- [Background] Köse D, Çınar N, Altınkaynak S. Yenidoğanın anne ve baba bağlanma süreci. STED Dergisi 2013; 226: 239-245.
- [Background] Menekşe ve Çınar N, Anne Bebek Bağlanması, İçinde Anne v eÇocuk Sağlığı İlk 1000 gün (Eds. Nursan Çınar, Sevil Şahin), Akademisyen Kitabevi,2020, 425-451.
- [Background] Mercer RT. Becoming a mother versus maternal role attainment. J Nurs Scholarsh. 2004;36(3):226-32. doi: 10.1111/j.1547-5069.2004.04042.x. PMID 15495491
- [Background] Nacar EH, Gökkaya F. Bağlanma ve maternal bağlanma konusunda bir derleme. Cyprus Turkish Journal of Psychiatry & Psychology 2019; 1 (1): 50-56.
- [Background] Pisoni C, Garofoli F, Baiardini I, Tzialla C, Stronati M. The development of parents-infant relationship in high-risk pregnancies and preterm birth. Journal of Pediatric and Neonatal Individualized Medicine 2014b;3 (2): 1-7.
- [Background] Scatliffe N, Casavant S, Vittner D, Cong X. Oxytocin and early parent-infant interactions: A systematic review. Int J Nurs Sci. 2019 Sep 12;6(4):445-453. doi: 10.1016/j.ijnss.2019.09.009. eCollection 2019 Oct 10. PMID 31728399